CLINICAL TRIAL: NCT04493242
Title: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles Infusion Treatment for COVID-19 Associated Acute Respiratory Distress Syndrome (ARDS): A Phase II Clinical Trial
Brief Title: Extracellular Vesicle Infusion Treatment for COVID-19 Associated ARDS
Acronym: EXIT-COVID19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Direct Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DB-EF-PHASEII-001
Expanded Access: NCT04657458 (No longer available)
Record Dates: First submitted 2020-07-29; First posted 2020-07-30 (Actual); Results first posted 2023-04-11 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; ARDS
Keywords: COVID-19; ARDS; Extracellular Vesicles; Exosome
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Multi-center, double-blinded, placebo-controlled, randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Normal saline 100 mL
  Interventions: Other: Intravenous normal saline
- Experimental Dose 1 (Experimental): Normal saline 90 mL and ExoFlo 10 mL
  Interventions: Biological: ExoFlo
- Experimental Dose 2 (Experimental): Normal saline 85 mL and ExoFlo 15 mL
  Interventions: Biological: ExoFlo

INTERVENTIONS:
Biological: ExoFlo — Intravenous administration of bone marrow mesenchymal stem cell derived extracellular vesicles
  Arms: Experimental Dose 1; Experimental Dose 2
Other: Intravenous normal saline — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of intravenous administration of bone marrow derived extracellular vesicles, ExoFlo, versus placebo as treatment for moderate-to-severe Acute Respiratory Distress Syndrome (ARDS) in patients with severe COVID-19.

DETAILED DESCRIPTION:
This is a Phase II, double-blinded, placebo-controlled, randomized controlled trial that enrolled 102 subjects that were admitted with COVID-19 associated moderate-to-severe ARDS across 6 sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (either by the individual or by the individual's healthcare proxy).
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18-85.
4. COVID-19 positive as defined by positive Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) SARS-CoV-2.
5. Moderate to severe ARDS as defined by modified Berlin definition, * which includes timing within 1 week of known clinical insult or new or worsening respiratory symptoms; bilateral opacities not fully explained by effusions, or lung collapse; respiratory failure not fully explained by cardiac failure or fluid overload; PaO2/FiO2 ≤ 200 mm Hg.

   *Modified Berlin definition used in this study is the full Berlin definition, albeit without the PEEP specification, which implies mechanical ventilation.
6. Hypoxia requiring noninvasive oxygen support such as Nasal Cannula (NC), Nonrebreather (NRB), Bilevel Positive Airway Pressure (BIPAP), Continuous Positive Airway Pressure (CPAP), high flow nasal cannula oxygen (HFNC O2) or mechanical ventilation (MV) despite initiating standard of care.
7. If the candidate is either a male or female of reproductive potential, he or she must agree to use of double barrier method of highly effective birth control contraception such as condoms with oral contraceptive pill or choose to remain abstinent if already practicing abstinence during the screening period. The required duration of usage of double barrier method OR maintenance of abstinence must include the time from the beginning of the screening period until 90 days following the last dose of the study treatment.

Exclusion Criteria:

1. Vulnerable populations such as pregnant patients, children, individuals with severe physical or mental disabilities who cannot provide meaningful consent.
2. Active malignancy requiring treatment within the last five years.
3. Major physical trauma in the last 5 days, including motor vehicle accidents, assaults, mechanical falls with sequelae of significant bleeding or craniofacial bruising, and surgeries.
4. Active tuberculosis or cystic fibrosis.
5. Severe chronic respiratory disease including chronic obstructive pulmonary disease or pulmonary fibrosis requiring home oxygen > 5L/min.
6. Use of extracorporeal membrane oxygenation (ECMO) during the current hospitalization.
7. Pre-existing pulmonary hypertension.
8. Severe pre-existing hepatic impairment (presence of cirrhosis, liver function tests (LFTs) ≥ 6x baseline, INR ≥ 2.0).
9. Pre-existing Chronic Kidney Disease (CKD) stage IIIb or End Stage Renal Disease (ESRD) prior to onset of COVID-19 (stage I, II, and IIIa are acceptable)
10. Irreversible coagulopathy (e.g., frequently occluded vascular access despite anticoagulation, precipitous platelet drops concurrent with end-organ damage suggesting consumptive process) or irreversible bleeding disorder (e.g., frequent bleeding from vascular access, endotracheal tubes, and foley).
11. Pneumonia clearly attributable to a non-COVID-19 related process, including aspiration pneumonia or pneumonia that is exclusively bacterial, or originating from a diagnosed alternative virus (e.g., influenza).
12. Patients who are not full code.
13. Endotracheal intubation duration ≤ 24 hours.
14. Moribund-expected survival < 24 hours.
15. Severe metabolic disturbances on presentation (e.g., ketoacidosis, pH < 7.3)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bill Arana, Study Director — Direct Biologics, LLC
Locations (6):
- United States (6):
  - Direct Biologics Investigational Site, Sheffield, Alabama
  - Direct Biologics Investigational Site, Anaheim, California
  - Direct Biologics Investigational Site, Sayre, Pennsylvania
  - Direct Biologics Investigational Site, Houston, Texas
  - Direct Biologics Investigational Site, Lubbock, Texas
  - Direct Biologics Investigational Site, Mesquite, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lightner AL, Sengupta V, Qian S, Ransom JT, Suzuki S, Park DJ, Melson TI, Williams BP, Walsh JJ, Awili M. Bone Marrow Mesenchymal Stem Cell-Derived Extracellular Vesicle Infusion for the Treatment of Respiratory Failure From COVID-19: A Randomized, Placebo-Controlled Dosing Clinical Trial. Chest. 2023 Dec;164(6):1444-1453. doi: 10.1016/j.chest.2023.06.024. Epub 2023 Jun 23. PMID 37356708
- See also: Direct Biologics, LLC — https://directbiologics.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 121 subjects were screened and 102 subjects were enrolled in the study at 6 investigative sites in the United States from 24 SEP 2020 to 22 MAY 2021.
Pre-assignment Details: Subjects that remained eligible per inclusion/exclusion criteria were randomized and equally distributed in the three study arms.
Period: Overall Study
Arm/Group | Experimental Dose 2 | Experimental Dose 1 | Placebo
Started | 34 | 34 | 34
Received 1 Dose Only | 7 | 5 | 7
Received 2 Doses | 27 | 29 | 27
Subjects Who Did Not Receive a Full Dose at Any Dose (Dose 1 or 2) | 1 | 0 | 0
Completed | 20 | 16 | 17
Not Completed | 14 | 18 | 17
Not completed — Death | 10 | 14 | 16
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Subjects Discharged from Hospital Prior to End of Study | 1 | 1 | 0
Not completed — Subjects Whose Status as of the End of Study Was Unknown | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set consisted of all participants who received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Dose 2 | Experimental Dose 1 | Placebo | Total
Number analyzed (Participants) | 34 | 34 | 34 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (14.97) | 62.1 (13.47) | 58.5 (11.76) | 59.1 (13.52)
Age, Customized [Count of Participants; unit: Participants]
  Age ≥ 65 | 8 | 14 | 10 | 32
  Age < 65 | 26 | 20 | 24 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 10 | 35
  Male | 22 | 21 | 24 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 4 | 10
  White | 21 | 31 | 26 | 78
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 3 | 8
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index- used to classify different weight types:
  Underweight: Less than 18.5 Optimum range: 18.5 to 24.9 Overweight: 25 to 29.9 Class I obesity: 30 to 34.9 Class II obesity: 35 to 39.9 Class III obesity: More than 40 Population: Unknown BMI for one subject in Experimental Dose 2 arm.
  kg/m^2
    number analyzed (Participants) | 33 | 34 | 34 | 101
    (all) | 34.98 (9.459) | 35.63 (10.939) | 34.24 (8.526) | 34.95 (9.615)
Respiratory Rate [Mean (Standard Deviation); unit: breaths/min] | 23.8 (5.38) | 24.4 (5.41) | 25.2 (7.90) | 24.5 (6.31)
Intubated Prior to Enrolling into the Study [Count of Participants; unit: Participants] | 2 | 1 | 4 | 7
Time from the First COVID-19 Diagnosis to the First IP Dose Date [Mean (Standard Deviation); unit: days] | 10.0 (6.55) | 9.1 (4.36) | 9.5 (4.12) | 9.5 (5.09)
Total SOFA Score [Mean (Standard Deviation); unit: scores on a scale] — Sequential Organ Failure Assessment Score- morbidity severity score and mortality estimation tool. The SOFA Score ranges from 0 to 24.
  SOFA Scores are used to estimate mortality risk. 0 to 6= <10% Mortality 7 to 9 = 15-20% Mortality 10 to 12= 40-50% Mortality 13 to 14= 50-60% Mortality 15= >80% Mortality 15 to 24= >90% Mortality Population: Unknown SOFA score for one subject in the placebo arm.
  scores on a scale
    number analyzed (Participants) | 34 | 34 | 33 | 101
    (all) | 3.2 (1.78) | 2.9 (1.20) | 3.2 (1.88) | 3.1 (1.64)
P/F Ratio [Mean (Standard Deviation); unit: mmHg] — Partial Pressure of Arterial Oxygen to Fraction of Inspired Oxygen Ratio Hypoxemia: mild (200 mm Hg < PaO2/FiO2 ≤ 300 mm Hg), moderate (100 mm Hg < PaO2/FiO2 ≤ 300 mm Hg), and severe (PaO2/FiO2 ≤ 100 mm Hg) Population: Unknown P/F Ratio data from 17 subjects in experimental dose 2, 15 subjects in experimental dose 1, and 16 subjects in placebo arms.
  mmHg
    number analyzed (Participants) | 17 | 19 | 18 | 54
    (all) | 115.202 (61.5299) | 113.824 (48.5386) | 102.952 (43.0002) | 110.634 (50.6610)
P/F Ratio [Count of Participants; unit: Participants]
  P/F Ratio < 100 mmHg | 10 | 9 | 10 | 29
  P/F Ratio ≥ 100 mmHg | 7 | 10 | 8 | 25
  Unknown P/F Ratio | 17 | 15 | 16 | 48
Prior Therapy [Count of Participants; unit: Participants] — Started prior to the first dose of IP regardless of its end date. Population: Measured for those subjects that started prior therapy prior to the first dose of IP.
  Participants
    Remdesivir: number analyzed (Participants) | 30 | 27 | 30 | 87
    Remdesivir | 17 | 21 | 23 | 61
    Convalescent Plasma: number analyzed (Participants) | 30 | 27 | 30 | 87
    Convalescent Plasma | 7 | 9 | 9 | 25
    Dexamethasone: number analyzed (Participants) | 30 | 27 | 30 | 87
    Dexamethasone | 26 | 25 | 27 | 78

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of 60-day Mortality Rate
Description: To evaluate the 60-day mortality rate for IP 15mL as a treatment for COVID-19 associated moderate to severe ARDS compared to placebo. Reducing the mortality rate for hospitalized patients with COVID-19 associated ARDS is a measure of the treatment effect.
Time Frame: 60 days
Population: The Intention to Treat Analysis set consisted of all participants who received study drug. The number of subjects who died within 60 days is captured in the Outcome Measure Data Table.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Dose 2 | Experimental Dose 1 | Placebo
Number analyzed (Participants) | 34 | 34 | 34
Participants | 10 | 14 | 16
Statistical Analysis 1: Comparison: Experimental Dose 2 vs Placebo; Test type: Other — log-rank test; p = 0.1343, Chi-squared

2. Secondary Outcome: Overall Survival Rates
Description: Reducing the mortality rate for hospitalized patients with COVID-19 associated ARDS is a measure of the treatment effect.
Time Frame: Days 15, 30, 60
Population: The Intention to Treat Analysis set consisted of all participants who received study drug.
Measure: Number; unit: Survival Percentage
Arm/Group | Experimental Dose 2 | Experimental Dose 1 | Placebo
Number analyzed (Participants) | 34 | 34 | 34
Survival Percentage
  Overall Survival Rate at 15 Days (Kaplan-Meier Method) | 78.8 | 77.8 | 75.8
  Overall Survival Rate at 30 Days (Kaplan-Meier Method) | 72.7 | 67.7 | 63.7
  Overall Survival Rate at 60 Days (Kaplan-Meier Method) | 69.6 | 53.4 | 51.6

3. Secondary Outcome: Proportion of Discharged Patients
Description: Discharge is an unbiased measure of overall clinical improvement.
Time Frame: Days 7, 30, 60
Population: The Intention to Treat Analysis Set consisted of all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Dose 2 | Experimental Dose 1 | Placebo
Number analyzed (Participants) | 34 | 34 | 34
Participants
  Subjects Who Discharged Within 7 Days | 11 | 9 | 11
  Subjects Who Discharged Within 30 Days | 19 | 17 | 17
  Subjects Who Discharged Within 60 Days | 20 | 18 | 17

4. Secondary Outcome: Time to Discharge
Description: Discharge is an unbiased measure of overall clinical improvement.
Time Frame: Number of days from the date of randomization until documented discharge from hospital, up to 60 days.
Population: Intention-to-Treat (ITT) Analysis set consists of all randomized patients. Patients were analyzed according to the randomized treatment arm.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Experimental Dose 2 | Experimental Dose 1 | Placebo
Number analyzed (Participants) | 34 | 34 | 34
days | 22 [6 to NA] — N/A: The upper 95% confidence interval cannot be estimated due to an insufficient number of discharged participants to estimate a standard error. | 29 [9 to NA] — N/A: The upper 95% confidence interval cannot be estimated due to an insufficient number of discharged participants to estimate a standard error. | NA [7 to NA] — Median was not reached due to an insufficient number of discharged patients. N/A: The upper 95% confidence interval cannot be estimated due to an insufficient number of discharged participants to estimate a standard error.

5. Secondary Outcome: Incidence of Treatment Emergent Serious Adverse Events
Description: Safety comparison performed between IP 15 mL and placebo arms
Time Frame: 61 days
Population: The Safety Analysis Set consisted of all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Dose 2 | Experimental Dose 1 | Placebo
Number analyzed (Participants) | 34 | 34 | 34
Participants
  Any TEAEs- Any Grade | 24 | 26 | 23
  Any TEAEs- Grade 3 or 4 | 5 | 9 | 5
  Serious TEAEs- Any Grade | 10 | 18 | 16
  Serious TEAEs- Grade 3 or 4 | 3 | 7 | 3
  Study Treatment-Related TEAEs | 0 | 0 | 1
  Study Treatment-Related Serious TEAEs | 0 | 0 | 0
  TEAEs That Led to Dose Interruption | 1 | 0 | 0
  TEAEs That Led to Missing Dose or Discontinued the Treatment Early | 0 | 0 | 1
  TEAEs That Led to Death | 10 | 13 | 16

6. Secondary Outcome: Ventilation Free Days
Description: Number of days for which patients are not on mechanical ventilation.
Time Frame: Within 60 days of follow-up
Population: The Intention to Treat Analysis set consisted of all participants who received study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Experimental Dose 2 | Experimental Dose 1 | Placebo
Number analyzed (Participants) | 34 | 34 | 34
days | 41.3 (25.78) | 32.0 (26.23) | 33.9 (28.06)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected within 60 days from the last dose.
Description: At each visit, the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Experimental Dose 2 | Experimental Dose 1 | Placebo
All-Cause Mortality (participants affected / at risk) | 10/34 | 14/34 | 16/34
Serious Adverse Events (participants affected / at risk) | 11/34 | 18/34 | 16/34
Other Adverse Events (participants affected / at risk) | 25/34 | 25/34 | 22/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Dose 2 (N=34) | Experimental Dose 1 (N=34) | Placebo (N=34)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Arteriospasm Coronary (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 2 (2) | 4 (4) | 4 (4)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Brain Injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain Oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Ischemia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 12 (12) | 9 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 6 (6)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral Ischemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Dose 2 (N=34) | Experimental Dose 1 (N=34) | Placebo (N=34)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2)
Anaemia Macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Hyponatraemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 5 (5) | 8 (8) | 8 (8)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 3 (3)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Blood Glucose Increased (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1)
Diabetes Mellitus (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Endocrine disorders) | 1 (1) | 3 (3) | 3 (3)
Type 2 Diabetes Mellitus (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Ophthalmic Herpes Zoster (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colonic Abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fall (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid Overload (General disorders) | 0 (0) | 2 (2) | 1 (1)
Generalised Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Hypocalcaemia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Hypoglycaemia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (General disorders) | 7 (7) | 8 (8) | 7 (7)
Hypophosphataemia (General disorders) | 0 (0) | 2 (2) | 4 (4)
Intensive Care Unit Acquired Weakness (General disorders) | 1 (1) | 0 (0) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 2 (2)
Vitamin D Deficiency (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary Disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice Cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candida Test Positive (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterococcal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Escherichia Coli (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Pneumonia Staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Fungal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection Enterococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Escherichia Test Positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Fibrin D Dimer Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Investigations) | 0 (0) | 4 (4) | 7 (7)
Hypernatraemia (Investigations) | 1 (1) | 1 (1) | 0 (0)
Hyperphosphataemia (Investigations) | 1 (1) | 1 (1) | 0 (0)
Klebsiella Test Positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver Function Test Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Morganella Test Positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas Test Positive (Investigations) | 0 (0) | 0 (0) | 2 (2)
Serratia Test Positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Stenotrophomonas Test Positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Troponin I Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Adjustment Disorder with Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 9 (9) | 4 (4)
Confusional State (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3)
Catheter Site Pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Endotracheal Intubation Complication (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Subcutaneous Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fungal Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Non-disclosure agreements with PIs in place. PIs cannot disclose data for approximately 10 years.

DOCUMENTS (2):
  • Study Protocol (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT04493242/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT04493242/SAP_001.pdf